CLINICAL TRIAL: NCT01925300
Title: A Randomized, Open-label, Repeated-dose, Crossover Study to Investigate the Pharmacokinetic Drug Interactions Between Bisoprolol and Rosuvastatin in Healthy Adult Volunteers
Brief Title: Pharmacokinetic Interactions of Bisoprolol and Rosuvastatin
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CJ_BCS_101
Record Dates: First submitted 2013-08-15; First posted 2013-08-19 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-12

CONDITIONS: Healthy
Keywords: Pharmacokinetics; Pharmacodynamics; Safety; Tolerability
MeSH Terms: interventions — Bisoprolol; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Concor 5mg(Bisoprolol hemifumarate 5mg) 2Tab, qd (Experimental): Single administration : 6 days, per oral
  Interventions: Drug: Concor 5mg(Bisoprolol hemifumarate 5mg) 2Tab
- Crestor 20mg(Rosuvastatin calcium 20.80mg) 1Tab, qd (Experimental): Single administration : 6 days, per oral
  Interventions: Drug: Crestor 20mg(Rosuvastatin calcium 20.80mg) 1Tab
- Concor 5mg 2T and Crestor 20 mg 1Tab, qd (Experimental): Combination administration : 6 days, per oral
  Interventions: Drug: Concor 5mg 2T and Crestor 20 mg 1Tab

INTERVENTIONS:
Drug: Concor 5mg(Bisoprolol hemifumarate 5mg) 2Tab
  Arms: Concor 5mg(Bisoprolol hemifumarate 5mg) 2Tab, qd
Drug: Crestor 20mg(Rosuvastatin calcium 20.80mg) 1Tab
  Arms: Crestor 20mg(Rosuvastatin calcium 20.80mg) 1Tab, qd
Drug: Concor 5mg 2T and Crestor 20 mg 1Tab
  Arms: Concor 5mg 2T and Crestor 20 mg 1Tab, qd

SUMMARY:
This study is designated to evaluate the pharmacokinetic interactions of bisoprolol and rosuvastatin in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Male volunteers in the age between 20 and 55 years old(inclusive)
* Body mass index (BMI) in the range of 18.5 to 27 kg/m2(inclusive)
* Medically healthy with no clinically significant vital signs (sitting position blood pressure, pulse rate) (90 mmHg ≤ systolic blood pressure ≤ 150 mmHg, 60 mmHg ≤ diastolic blood pressure ≤ 100 mmHg, 50 beats per minute ≤ pulse rate ≤ 100 beats per minute)
* Available for the entire study period
* Understand the requirements of the study and voluntarily consent to participate in the study

Exclusion Criteria:

* Subjects with a history of gastrointestinal diseases which might significantly change ADME(Absorption, Distribution, Metabolism and Excretion) of medicines
* History of clinically significant arrhythmic, peripheral vascular,thyroid, bronchospasm, asthma disease
* Subjects with anaphylaxis to bisoprolol and/or rosuvastatin
* History of drug abuse
* History of caffeine, alcohol, smoking abuse

  * caffeine(coffee,tea,coke) or grapefruit juice > 4cups/day
  * smoking > 20 cigarettes/day
  * alcohol > 140g/week
* Clinical laboratory test values are outside the accepted normal range

  * AST(Aspartate Transaminase), ALT(ALanine Transaminase)( > 1.5 times to normal range
  * CK(Creatine Kinase) > 1.5 times to normal range
  * Estimated GFR(Glomerular Filtration Rate) < 60 mL/min
* Subjects with whole blood donation within 60days, component blood donation within 30days and blood transfusion within 30days prior to study medication dosing
* Subjects considered as unsuitable based on medical judgement by investigators

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-07; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Assessment of the drug-drug interactions of bisoprolol and rosuvastatin: Cmax,ss(Maximum steady-state plasma drug concentration during a dosage interval ), AUCτ(Area Under the Curve) | 6 days
  Administration of Investigational Product : 6 days/period(total 3 period)

SECONDARY OUTCOMES:
Assessment of the bisoprolol and rosuvastatin:tmax,ss(Time to reach Cmax,ss), t1/2, Cmin,ss(Minimum steady-state plasma drug concentration during a dosage interval ), CL/Fss(Oral Clearance), Vd/Fss(Apparent Volume of Distribution) | 6 days
  Administration of Investigational Product : 6 days/period(total 3 period)

CONTACTS AND LOCATIONS:
Overall Officials: Jae-wook Ko, phD, Principal Investigator — Samsung Medical Conter